CLINICAL TRIAL: NCT06228378
Title: Comparative Spectroscopic Analysis of Synovial Fluid From the Stable and Unstable Ankle
Acronym: ALSACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01300-43
Record Dates: First submitted 2023-12-14; First posted 2024-01-29 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, open-label study of patients undergoing ankle stabilisation surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unstable ankle (Experimental): Unstable ankle
  Interventions: Other: Raman microspectroscopy
- Stable ankle (Active Comparator)
  Interventions: Other: Raman microspectroscopy

INTERVENTIONS:
Other: Raman microspectroscopy — Raman microspectroscopy is a non-destructive method for observing and characterising the molecular composition and external structure of a biological sample based on the phenomenon of inelastic light scattering (Raman effect).

SUMMARY:
A population of patients with chronic ankle instability for whom arthroscopic ligament stabilisation was indicated.

Main objective: to use the Raman microspectroscopy technique to characterise the synovial fluid of the unstable ankle in comparison with the synovial fluid of the healthy ankle.

DETAILED DESCRIPTION:
Single-centre, prospective, open-label study of patients undergoing ankle stabilisation surgery.

Patients will participate in the study for six months. Three arthrocentheses with synovial fluid sampling will be performed Two at D0: on the healthy ankle and the pathological ankle One at M6: on the operated ankle A follow-up visit will take place 10 days after the arthrocentesis performed at D0 and after the one performed at M6. The purpose of these visits, which are carried out systematically by the centre's doctors as part of the surgical procedures, is to check that there are no complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over who have signed their consent to participate in the study
* Patients with chronic unilateral lateral ankle instability
* Patients who have not responded to medical treatment and for whom arthroscopic stabilisation of the ankle is planned.

Exclusion Criteria:

* Any history, anomaly or symptom relating to the contralateral ankle
* Patient under court protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Spectral intensity of synovial fluid components | Month 6
  Spectral intensity of synovial fluid components :
  Raman microspectroscopy is a non-destructive method for observing and characterising the molecular composition and external structure of a biological sample based on the phenomenon of inelastic light scattering.
  Four regions of interest (ROIs) are defined at the four cardinal points in the peripheral zone where the pre-concentration of solutes is maximal. Six points are mapped in each ROI. Each drop is thus defined by 4 x 6 points, making it possible to check intra- and inter-ROI homogeneity. Spectral acquisitions were carried out after illumination by a laser source.
  The mean spectrum of each LS drop is defined as the average of the four mean spectra of the ROIs, originating from the four cardinal points of the drop. The component Raman bands are identified and assigned on the basis of bibliographic data.

SECONDARY OUTCOMES:
Functional criterion (American Orthopaedic Foot and Ankle Society-AOFAS score) | Month 6
  Functional criterion (AOFAS score)
Tribological criteria (drop surface measurement) | Month 6
  Tribological criteria (drop surface measurement)
Tribological criteria (drop thickness measurement) | Month 6
  Tribological criteria (drop thickness measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre HARDY, MD, Principal Investigator — Clinique du sport
Locations (1):
- Clinique du Sport, Paris, France